CLINICAL TRIAL: NCT06943664
Title: Phase II Trial: Photoimmunotherapy and Anti-PD1 in Patients With Refractory Inoperable and Metastatic Non-Small Cell Lung Cancer
Brief Title: Photoimmunotherapy With ASP-1929 and Cemiplimab for the Treatment of Refractory, Inoperable, and Metastatic Stage IIIB-IV Non-small Cell Lung Cancer
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Roswell Park Cancer Institute (Other)
Collaborators: Rakuten Medical, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: I-3845023; NCI-2025-02417 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); I-3845023 (Other: Roswell Park Cancer Institute)
Record Dates: First submitted 2025-04-17; First posted 2025-04-24 (Actual); Last update posted 2025-12-15 (Actual); Status verified 2025-12

CONDITIONS: Lung Non-Small Cell Carcinoma; Metastatic Lung Non-Small Cell Carcinoma; Refractory Lung Non-Small Cell Carcinoma; Stage IIIB Lung Cancer AJCC v8; Stage IIIC Lung Cancer AJCC v8; Stage IV Lung Cancer AJCC v8
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Lung Neoplasms | interventions — Specimen Handling; cemiplimab; Magnetic Resonance Spectroscopy; Photochemotherapy; Thoracic Surgery, Video-Assisted

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Treatment (photoimmunotherapy, ASP-1929, cemiplimab) (Experimental): Patients receive cemiplimab IV over 30 minutes on days 1, 22, and 43 of each cycle and ASP-1929 IV over 2 hours on day 8 of each cycle. Patients undergo EB-PIT via standard of care VATS once on day 9 of cycle 1 or I-PIT via EBUS or robotic bronchoscopy up to 3 times on day 9 of cycles 1, 2, and/or 3. Cycles repeat every 9 weeks for up to 2 years in the absence of disease progression or unacceptable toxicity. Additionally, patients undergo blood sample collection, CT and/or PET/CT or MRI throughout the study.
  Interventions: Procedure: Biospecimen Collection; Biological: Cemiplimab; Biological: Cetuximab Sarotalocan Sodium; Procedure: Computed Tomography; Other: Electronic Health Record Review; Procedure: Endobronchial Ultrasound Bronchoscopy; Procedure: Magnetic Resonance Imaging; Procedure: Photoimmunotherapy; Procedure: Positron Emission Tomography; Procedure: Robotic Bronchoscopy; Procedure: Video-Assisted Thoracic Surgery

INTERVENTIONS:
Procedure: Biospecimen Collection — Undergo blood sample collection
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Biological: Cemiplimab — Given IV
  Other Names: Cemiplimab RWLC; Cemiplimab-rwlc; Libtayo; REGN 2810; REGN-2810; REGN2810
Biological: Cetuximab Sarotalocan Sodium — Given IV
  Other Names: ASP 1929; ASP-1929; ASP1929; Cet-IR700; Cetuximab-IR700 Conjugate RM-1929; RM-1929
Procedure: Computed Tomography — Undergo CT or PET/CT
  Other Names: CAT; CAT Scan; Computed Axial Tomography; Computerized Axial Tomography; Computerized axial tomography (procedure); Computerized Tomography; Computerized Tomography (CT) scan; CT; CT Scan; tomography
Other: Electronic Health Record Review — Ancillary studies
Procedure: Endobronchial Ultrasound Bronchoscopy — Undergo EBUS
  Other Names: EBUS; Endobronchial Ultrasound
Procedure: Magnetic Resonance Imaging — Undergo MRI
  Other Names: Magnetic Resonance; Magnetic Resonance Imaging (MRI); Magnetic resonance imaging (procedure); Magnetic Resonance Imaging Scan; Medical Imaging, Magnetic Resonance / Nuclear Magnetic Resonance; MR; MR Imaging; MRI; MRI Scan; MRIs; NMR Imaging; NMRI; Nuclear Magnetic Resonance Imaging; sMRI; Structural MRI
Procedure: Photoimmunotherapy — Undergo EB-PIT
  Other Names: Photodynamic Light Therapy
Procedure: Photoimmunotherapy — Undergo I-PIT
  Other Names: Photodynamic Light Therapy
Procedure: Positron Emission Tomography — Undergo PET/CT
  Other Names: Medical Imaging, Positron Emission Tomography; PET; PET Scan; Positron emission tomography (procedure); Positron Emission Tomography Scan; Positron-Emission Tomography; PT
Procedure: Robotic Bronchoscopy — Undergo robotic bronchoscopy
  Other Names: Robot-Assisted Bronchoscopy; Robotic-Assisted Bronchoscopy
Procedure: Video-Assisted Thoracic Surgery — Undergo VATS
  Other Names: VATS; Video-Assisted Thoroscopic Surgery

SUMMARY:
This phase II trial tests how well photoimmunotherapy (PIT) with ASP-1929 in combination with cemiplimab works in treating patients with stage IIIB-IV non-small cell lung cancer (NSCLC) that has not responded to previous treatment (refractory), that is not suitable for surgery (inoperable), or that has spread from where it first started to other places in the body (metastatic). PIT is a treatment that combines drugs that become active when exposed to light, such as ASP-1929, with immunotherapy to target and kill tumor cells. ASP-1929 combines cetuximab with a light-sensitive component, sarotalocan. Cetuximab is in a class of medications called monoclonal antibodies. It binds to a protein called epidermal growth factor receptor (EGFR), which is found on some types of tumor cells. This may help keep tumor cells from growing. Sarotalocan is a fluorescent dye, infrared-activated fluorescent dye 700, that is light sensitive, and when activated by a special type of laser light, helps destroy or change tumor cells. Immunotherapy with monoclonal antibodies, such as cemiplimab, may help the body's immune system attack the tumor, and may interfere with the ability of tumor cells to grow and spread. Giving PIT with ASP-1929 in combination with cemiplimab may kill more tumor cells in patients with refractory, inoperable, or metastatic stage IIIB-IV NSCLC.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To assess objective response rate of tumors and lymph nodes following photoimmunotherapy and anti-PD1.

SECONDARY OBJECTIVES:

I. Overall survival following photoimmunotherapy and anti-PD1. II. To assess median progression free survival following photoimmunotherapy and anti-PD1.

III. To assess the relationship between light irradiance and fluence dose volume histograms and objective tumors response following photoimmunotherapy and anti-PD1.

IV. To evaluate the safety of cetuximab sarotalocan sodium (ASP-1929) photoimmunotherapy in combination with immune checkpoint inhibitors in patients with refractory inoperable and metastatic non-small cell lung cancer.

EXPLORATORY OBJECTIVES:

I. To assess the relationship between changes of circulating tumor deoxyribonucleic acid (DNA) (ctDNA) levels and objective response of tumors.

II. To assess the relationship between levels of EGFR expression and the objective response of tumors.

OUTLINE:

Patients receive cemiplimab intravenously (IV) over 30 minutes on days 1, 22, and 43 of each cycle and ASP-1929 IV over 2 hours on day 8 of each cycle. Patients undergo external beam (EB)-PIT via standard of care video-assisted thoracic surgery (VATS) once on day 9 of cycle 1 or interstitial (I)-PIT via endobronchial ultrasound (EBUS) or robotic bronchoscopy up to 3 times on day 9 of cycles 1, 2, and/or 3. Cycles repeat every 9 weeks for up to 2 years in the absence of disease progression or unacceptable toxicity. Additionally, patients undergo blood sample collection, computed tomography (CT) and/or positron emission tomography (PET)/CT or magnetic resonance imaging (MRI) throughout the study.

After completion of study treatment, patients are followed up every 3 months for up to 2 years.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years of age
* Have an Eastern Cooperative Oncology Group (ECOG) performance status of 0-2
* Subjects with histologically or cytologically confirmed stage IIIB-IV NSCLC
* Subjects lacking actionable genetic mutations must have been previously treated with (a) anti-PD-1/PD-L1 therapy; and (b) platinum-based chemotherapy, either as combination or sequentially for metastatic disease and have progressed on or after therapy. Individuals who cannot tolerate or have previously refused platinum-based chemotherapy or who are unable to receive it are eligible to enroll based on progression after anti-PD-1/PD-L1 therapy alone
* NSCLC with known actionable genomic alteration (e.g., EGFR, ALK, ROS1, BRAF) must have received all approved targeted therapies and have progressed (data capture not necessary for ALK, ROS1, BRAF)
* Subjects have at least two lesions of measurable disease by Response Evaluation Criteria in Solid Tumors (RECIST) 1.1
* At least one site of disease accessible to photoimmunotherapy. Thus, the therapeutic 690-nm laser light can be administered via insertion of optical fiber/s in the target tumor for interstitial photoimmunotherapy (I-PIT), or target tumors can be illuminated with external beam photoimmunotherapy (EB-PIT)
* Absolute neutrophil count: ≥ 1,000/µL
* Platelets: ≥ 100,000/µL
* Total bilirubin: ≤ institutional upper limit of normal (ULN)
* Aspartate aminotransferase (AST)(serum glutamic oxaloacetic transaminase [SGOT])/alanine aminotransferase (ALT)(serum glutamic pyruvic transaminase [SGPT]): ≤ 3 x institutional ULN
* Creatinine clearance (CrCl) ≥ 50 mL/min (Cockcroft-Gault)
* Patient has not received a transfusion within 2 weeks prior to screening
* Female patients of childbearing potential must have a negative pregnancy test at screening and must be willing to use 2 methods of highly effective birth control while on study or be surgically sterile, or abstain from heterosexual sexual activity for the course of the study through 120 days after the last dose of anti-PD1 treatment. Should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately
* Male participants must agree to use a highly effective method of contraception starting with the first dose of study medication through 120 days after the last dose of anti-PD1 treatment
* Participant must understand the investigational nature of this study and sign an independent ethics committee/institutional review board approved written informed consent form prior to receiving any study related procedures

Exclusion Criteria:

* Has received an investigational agent within 30 days prior to initial treatment or less than 4 half-lives of a previous drug
* Had a major surgery, (e.g., requiring general anesthesia) within 4 weeks before the first dose of study treatment or, will not have fully recovered from surgery prior to the first dose
* Patients who received chemotherapy or chemoimmunotherapy within 21 days or those who have not recovered from reversible adverse events prior to the scheduled surgery and interstitial or intraoperative PIT
* The participants received high dose or curative radiotherapy to the target tumor/s within 30 days prior to the planned I-PIT or EB-PIT
* Toxicity related to prior anticancer therapy that has not returned to grade ≤ 1 or baseline levels (except for alopecia, vitiligo, grade ≤ 2 peripheral neuropathy, and endocrinopathies that are stable on hormone replacement, which may be grade 2)
* History of immune-related adverse events (irAEs) from prior anticancer therapy leading to permanent treatment discontinuation
* History of solid organ or hematologic stem cell transplantation
* Prolonged corrected QT interval by Fredericia (QTcF) > 470 msec or clinically significant cardiac arrhythmia or electrophysiologic disease (e.g., placement of implantable cardioverter defibrillator or atrial fibrillation with uncontrolled rate or abnormalities in conduction or morphology of electrocardiogram [ECG] [e.g., complete left bundle branch block, third- or second-degree heart block, PR interval > 250 msec]). Note: Participants with cardiac pacemakers who are clinically stable are eligible
* Clinically significant cardiovascular disease, including any of the following within 6 months prior to signature of informed consent:

  * Myocardial infarction, severe or unstable angina, or coronary artery bypass surgery
  * Clinically significant arrhythmias (e.g., ventricular arrhythmias or atrial fibrillation with uncontrolled heart rate)
  * Congestive heart failure (New York Heart Association [NYHA] class III/IV)
  * Cerebrovascular accident, transient ischemic attack, or other arterial thromboembolic event
  * Myocarditis
* Active bleeding diathesis or requirement for therapeutic anticoagulation that cannot be interrupted or altered for procedures
* Patients with untreated or symptomatically unstable treated brain metastases or history of leptomeningeal disease should be excluded from this clinical trial because of their poor prognosis and because they often develop progressive neurologic dysfunction that would confound the evaluation of neurologic and other adverse events. Patients with treated and stable brain metastases (at least 28 days from last radiotherapy treatment) are eligible as long as steroids are not required for symptom management
* Known history of hepatitis B, hepatitis C or human immunodeficiency virus (HIV). Exceptions include past or resolved hepatitis B (defined as the presence of hepatitis B core antibody [anti-HBc] and absence of hepatitis B virus surface antigen [HBsAg]) and patients positive for hepatitis C (hepatitis C virus [HCV]) antibody if polymerase chain reaction is negative for HCV ribonucleic acid (RNA). HIV testing is not required in absence of clinical suspicion of HIV
* History of, or active autoimmune disorder, requiring systemic steroids or immunosuppressive agents. Exceptions allowed: Patients with autoimmune dermatologic conditions not requiring systemic steroids or immunosuppressive agents (e.g. vitiligo, eczema, etc.), endocrine-related autoimmune conditions receiving appropriate hormonal supplementation

  * Use of immunosuppressant drugs such as steroids, azathioprine, tacrolimus, cyclosporine, etc. is not permitted within 4 weeks before recruitment (exception allowed is use of steroids as hormone replacement therapy or as supportive medication e.g. anti-emesis, contrast allergy, pre-medication, etc. or other short-course therapy less than 2 weeks continuously within 4 weeks of study treatment)
* History of significant (≥ grade 3) cetuximab infusion reactions
* Evidence of interstitial lung disease or current active, noninfectious pneumonitis
* Active or prior documented autoimmune or inflammatory disorders (including inflammatory bowel disease [e.g. colitis or Crohn's disease], systemic lupus erythematosus, sarcoidosis syndrome, or Wegener syndrome [granulomatosis with polyangiitis, Graves' disease, rheumatoid arthritis, hypophysitis, uveitis, etc.]). The following are exceptions to this criterion:

  * Patients with vitiligo or alopecia
  * Patients with hypothyroidism (e.g. following Hashimoto syndrome) stable on hormone replacement
  * Any chronic skin condition that does not require systemic therapy
  * Patients without active disease in the last 5 years may be included
  * Patients with celiac disease controlled by diet alone
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements
* Any condition which in the investigator's opinion deems the participant an unsuitable candidate to receive ASP-1929
* Any condition which in the investigator's opinion deems the subject an unsuitable candidate to receive the experimental PIT or immunotherapy
* Pregnant or nursing female participants
* Unwilling or unable to follow protocol requirements

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Estimated)
Dates: Start 2026-01-15 (Estimated); Primary Completion 2027-05-01 (Estimated); Study Completion 2028-05-01 (Estimated)

PRIMARY OUTCOMES:
Overall response rate | Up to 2 years
  Will be defined as the proportion of patients who have a partial or complete response to therapy and will be assessed according to immune-modified Response Evaluation Criteria in Solid Tumors (RECIST) version (v) 1.1.

SECONDARY OUTCOMES:
Overall survival | From the treatment to time of death from any reason, assessed up to 2 years
  Will be defined as the time the patient is alive without tumor progression after treatment according to RECIST v 1.1. Will be estimated using the Kaplan-Meier estimator.
Median progression free survival (PFS) | Up to 2 years
  Will be defined as the time the patient is alive without tumor progression after treatment according to RECIST v 1.1. Will be estimated using the Kaplan-Meier estimator. Corresponding median PFS will be estimated along with the respective 95% confidence interval.
Relationship between the light irradiance and fluence in the photoimmunotherapy treated tumor and the objective response of treated and untreated tumors | Up to 2 years
  Will be determined by computing the dose volume histogram of the irradiance and fluence in the illuminated tumor/s and measuring the objective tumor response according to RECIST v 1.1. Will be analyzed using multivariate and univariate mixed effects logistic and standard logistic regression modeling.
Incidence of adverse events | From the first day of the administration of the ASP-1929 up to 30 days after last treatment of ASP-1929 with cemiplimab
  Will be evaluated in accordance with Common Terminology Criteria for Adverse Events v 5.0.

CONTACTS AND LOCATIONS:
Overall Officials: Prantesh Jain, Principal Investigator — Roswell Park Cancer Institute
Locations (1):
- Roswell Park Cancer Institute, Buffalo, New York, United States